CLINICAL TRIAL: NCT04700371
Title: Flexion-Induced Vessel Deformations and Restenosis After Stenting of the Popliteal Artery
Brief Title: Vessel Deformations and Restenosis After Stenting of the Popliteal Artery
Acronym: FIRESTEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support.
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Aljoscha Rastan, MD, Head of Endovascular Therapy, Angiology, Kantonsspital Aarau, Kantonsspital Aarau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0-2020
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease; Popliteal Artery Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interwoven stent (Active Comparator): Use of an interwoven nitinol stent to treat patients with arteriosclerotic lesions of the distal portion of the superficial artery and/or the popliteal artery.
  Interventions: Device: Interwoven stent
- Laser-cut stent (Active Comparator): Use of a laser-cut nitinol stent to treat patients with arteriosclerotic lesions of the distal portion of the superficial artery and/or the popliteal artery.
  Interventions: Device: Laser-cut stent

INTERVENTIONS:
Device: Interwoven stent — Interwoven nitinol stent placement in patients with arteriosclerotic lesions of the distal portion of the superficial artery and/or the popliteal artery.
  Arms: Interwoven stent
Device: Laser-cut stent — Laser-cut nitinol stent placement in patients with arteriosclerotic lesions of the distal portion of the superficial artery and/or the popliteal artery.
  Arms: Laser-cut stent

SUMMARY:
The femoro-popliteal (FP) artery is the most frequently treated vascular segment in patients with symptomatic peripheral artery disease (PAD), for which endovascular therapy became an established treatment option during the last decades. However, loss of primary patency and consecutive clinically driven target lesion revascularization (TLR) limit this procedure. Moreover, in the popliteal artery (PA), evidence about the best treatment strategy to prevent loss of patency and TLR is limited to only a few randomized controlled trials (RCT). Arterial deformations of the PA with its unique anatomical properties during leg flexion might explain the poor technical and clinical outcomes in this segment. Generally, a "leave nothing behind" strategy in the PA is preferred, but cannot be avoided in all cases due to e.g. flow limiting dissections or re-coil after balloon angioplasty. Basically two different self-expandable nitinol-based stent designs are available on the market. An interwoven nitinol and laser-cut nitinol stent. The interwoven nitinol stent has a higher radial force in comparison to the laser-cut stent and reveals higher patency rates in the FP arteries. However, a head-to-head comparison of these stents is missing and it remains unknown in which way different stent designs affect the deformation and hemodynamic behaviors of the PA during knee flexion.

DETAILED DESCRIPTION:
Randomized trial to investigate the impact of different stent designs on the target lesion restenosis rate in femoro-popliteal arteries. Immediately after stent implantation, sets of three orthogonal angiographic views (separated by an angle of > 25°) of the stented region (TL) will be obtained with the leg in supine position. This will be followed by intra-arterial imaging using Optical Coherence Tomography (OCT). OCT images (one pullback if the lesion length is < 75 mm, 2 pullbacks otherwise) of the TL will be acquired using the Dragonfly catheter. In addition, duplex ultrasound (DU) of the TL will be performed, including the arterial segments 10cm at proximal and distal edge of the TL. Thereafter, a bending cast will be used to obtain a knee/hip flexion of approximately 70°/20°. In this position the angiographic, OCT, and DU measurements will be repeated.

The OCT images will provide the shapes of the arterial lumen which will be used to generate 3D surface models (in .stl format). The X-ray images will be utilized to construct the 3D arterial centerline for the supine and flexed leg positions. These arterial centerlines will be used to quantify the axial deformation (in mm), twisting (in °), and curvature changes (in mm-1) along the length of the investigated segment. Additionally, the lumen profiles obtained from OCT images will be used to accurately estimate the radial deformations (in mm) in the lumen and define instances of arterial pinching during leg flexion (as the difference in lumen diameters between straight and flexed leg positions).

The geometries of the arterial lumens will be combined with their corresponding 3D arterial centerlines to generate patient-specific arterial models. Along with patient-specific boundary conditions obtained from DU measurements, these models will be transferred to a commercial software, to perform Computational Fluid Dynamics analyses. The changes in these parameters due to leg flexion, as well as due to different stent designs, will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study procedure,
* Presence of PAD (2 - 3 Rutherford-Becker class),
* Atherosclerotic de-novo lesion (stenosis >70% or occlusion) of the distal part of the superficial femoral artery and/or any part of the popliteal artery,
* Target lesion-length: 4cm to 12cm,
* Target vessel diameter: 5mm to 7mm,
* Guidewire must cross target lesion and located intraluminally before randomization,
* At least one (1) patent below-the knee artery (=with no stenosis >50%),
* Possibility to treat the target lesion with one (1) study stent
* Interventions in TASC A and B lesions to restore adequate blood flow, in the same index procedure, are allowed. This intervention must be prior to the treatment of the study lesion(s) and successful.

Exclusion Criteria:

* Pregnancy,
* Angiographic evidence of thrombus within the target lesion,
* Patients with acute critical limb ischemia (Rutherford-Becker class 4-6),
* Restenosis of the target lesion,
* Non-atherosclerotic obstructions of the target lesion,
* Aneurysm of the target lesion,
* Renal failure, defined as GFR, <40 mL/min/1.73m2,
* Patient's inability to follow the study procedures e.g. psychological disorders, dementia, etc.,
* Previous enrolment into an ongoing study,
* Known or suspected allergies or contraindications to aspirin and/or clopidogrel, heparin,
* Coagulation disorders, or general refusal of the patient to receive blood transfusions,
* Contrast allergy that cannot be treated,
* Thrombolysis therapy including 72 hours before the planned index procedure,
* Myocardial infarction or stroke <30 days prior to index procedure.
* Equipment is unavailable to fulfill study treatments.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 1 year post index procedure
  Primary patency of the target lesion measured by duplex ultrasound

SECONDARY OUTCOMES:
Changes in arterial flow within the target lesion | 6 weeks, 6 months, and 1 year post index procedure
  Changes in blood flow/hemodynamics caused by the different stent designs measured by Computational Fluid Dynamics

CONTACTS AND LOCATIONS:
Overall Officials: Aljoscha Rastan, Principal Investigator — Kantonsspital Aarau

IPD SHARING:
Plan to Share IPD: No